CLINICAL TRIAL: NCT05192668
Title: The Setting and Effect Evaluation of Quiet Time in Neonatal Intensive Care Unit
Brief Title: The Setting and Effect Evaluation of QT in NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: [2021]296
Record Dates: First submitted 2021-12-27; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Very Low Birth Weight Infant
Keywords: Quiet Time; Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quiet time care (Experimental): Reduce noise and centralize medical or nursing operations in the NICU
  Interventions: Other: Quiet time care
- Routine nursing care (No Intervention): Perform routine nursing care for the VLBWIs in the NICU

INTERVENTIONS:
Other: Quiet time care — This study is a non-self before and after control study. The data of VLBWIs in the control group is collected in the early stage, and the quiet time intervention is carried out in the later period, and the data of VLBWIs in the intervention group is collected
  Arms: Quiet time care

SUMMARY:
In order to create a better environment for growth and development for very low birth weight infants(VLBWIs), investigators introduce quiet time, which is an intervention method that reduces environmental noise in the ward and centralizes medical and nursing operations. By analyzing the weight gain of VLBWIs in the intervention group and the control group during hospitalization, the effect of setting a quiet time in the NICU on improving the growth and development of VLBWIs is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <1500g;
* Admit within 24 hours of birth;
* The guardian signs the informed consent.

Exclusion Criteria:

* Newborn with severe congenital malformations or various chromosomal diseases, genetic metabolic diseases, severe neurological diseases;
* Newborn who do not achieve discharge or death at the end of the study period.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mean weekly gain in weight of VLBWIs | From the day the VLBWI admitted to the day VLBWI discharged, about two months.
  The average weekly gain in weight of VLBWIs in the intervention group minus the average weekly gain in weight of VLBWIs in the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China